CLINICAL TRIAL: NCT00094003
Title: A Phase I, Open-Label, Dose Escalation Study of Intravenously Administered NS-9 in Subjects With Liver Metastases From Various Primary Cancers
Brief Title: Study of NS-9 in Patients With Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NS Pharma, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS9001
Record Dates: First submitted 2004-10-08; First posted 2004-10-11 (Estimated); Last update posted 2005-11-11 (Estimated); Status verified 2005-11

CONDITIONS: Liver Neoplasms; Neoplasm Metastasis; Local Neoplasm Recurrences
Keywords: Liver metastases; Colorectal cancer; Gastric cancer; Esophagus cancer; Breast cancer; Lung cancer; Skin cancer; Renal Cancer; Liver metastasis
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Neoplasm Recurrence, Local; Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Breast Neoplasms; Lung Neoplasms; Skin Neoplasms; Kidney Neoplasms | interventions — Poly I-C

INTERVENTIONS:
Drug: NS-9 [Poly I: Poly C]

SUMMARY:
This study is to investigate the safety of NS-9 and to see how well it is tolerated in patients with cancer that has metastasized (spread) to the liver from another primary tumor. NS-9 is a drug developed to go to the liver to cause cell death specifically in tumor cells. This study is also set up to determine the best dose to use.

DETAILED DESCRIPTION:
This study requires subjects to undergo 2 treatment cycles of NS-9. Each cycle consists of once daily, 1-hour I.V. infusions of the drug for 5 days followed by a 23-day rest period. During the rest period, subjects are seen at the clinic once weekly for evaluation. Subjects having favorable or stable results after 2 cycles may continue to receive NS-9 in the extension phase of the study until the disease progresses or until they get a side effect that prevents them from continuing with therapy.

After each two cycles, if appropriate, the liver tumor will be measured by radiologic imaging to compare it to its pre-treatment size.

ELIGIBILITY:
Inclusion Criteria:

* Male and female at least 18 years of age.
* Patients with liver metastases from various primary cancers for which no other curative treatment options exist.
* At least one measurable lesion (by CT or MRI)
* Life expectancy > 3 months
* Child-bearing potential women must have a negative serum pregnancy test
* ECOG performance status: 0-1
* Fully recovered from any previous cancer therapy or infection (at least 4 weeks from radiation or chemotherapy, at least 3 weeks from a major surgical procedure and at least 2 weeks from an exploration/biopsy)
* Discontinued from any other investigational drug for at least 30 days
* Serum calcium <11 mg/dL
* Absolute neutrophil count (ANC) ≥1,500/mm3, without growth factor support
* Hemoglobin ≥9.0 g/dL
* Platelet count ≥100,000/mm3
* Serum creatinine ≤1.5 times the upper limit of normal (ULN)
* Bilirubin ≤1.5 times ULN
* ALT and AST ≤3 times ULN
* Amylase and lipase ≤ ULN
* PT and PTT < 1.5 times ULN
* ECG with no acute abnormalities
* Afebrile (≤37.5C or 99.5F)
* Willingness and ability to comply with all study requirements

Exclusion Criteria:

* Subject is mentally or legally incapacitated, or has significant emotional or psychiatric problems.
* Concomitant primary malignant and/or non-malignant liver disease (primary liver cancer, acute or chronic hepatitis, cirrhosis, alcoholic liver disease).
* History of pancreatic disease (e.g., pancreatitis, pancreatic malignancy).
* New York Heart Association classification Class III or IV
* Uncontrolled intercurrent illnesses including but not limited to: hypertension, seizure disorder, renal, gastrointestinal, or hematological diseases.
* Clinically relevant systemic disease (other than the malignancy and malignancy-related hepatic dysfunction) making implementation of the protocol or interpretation of the study results difficult.
* Pregnant or nursing, or unwilling to or will not agree to use an effective and reliable contraceptive measure.
* Subject has received radiation to >25% of the total bone marrow.
* Subject has a history of any other illness that would preclude study participation.
* Subject has brain metastases.
* Subject has allergy to egg yolk.
* Subject receiving low-molecular weight heparin for treatment of a blood coagulation disorder (e.g., deep vein thrombosis, pulmonary embolism).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-09

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - MD Anderson Cancer Center, Houston, Texas